CLINICAL TRIAL: NCT03074695
Title: A Randomized Controlled Trial for Epidural Labor Analgesia: Comparison of Dural Puncture Epidural With Standard Labor Epidural Techniques
Brief Title: DPE Technique in Labor Epidural for Morbidly Obese Women
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pro00079368
Record Dates: First submitted 2017-02-16; First posted 2017-03-09 (Actual); Results first posted 2022-06-01 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Morbid Obesity; Labor Pain
MeSH Terms: conditions — Obesity, Morbid; Labor Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Dural Puncture Epidural (DPE) (Experimental): Women who have analgesia initiated with a DPE technique
  Interventions: Procedure: Dural puncture epidural (DPE); Drug: Dural puncture epidural (DPE)
- Standard Epidural (EPL) (Experimental): Women who have analgesia initiated with an epidural technique
  Interventions: Procedure: Standard Epidural (EPL); Drug: Standard Epidural (EPL)

INTERVENTIONS:
Procedure: Dural puncture epidural (DPE) — Epidural with spinal needle placed to confirm cerebral spinal fluid (CSF) position. No intrathecal dosing
  Arms: Dural Puncture Epidural (DPE)
Procedure: Standard Epidural (EPL) — Standard epidural placement
  Arms: Standard Epidural (EPL)
Drug: Dural puncture epidural (DPE) — Epidural with spinal needle placed to confirm CSF position. No intrathecal dosing. Ropivacaine 0.1% and Fentanyl 2mcg/mL.
  Arms: Dural Puncture Epidural (DPE)
Drug: Standard Epidural (EPL) — Standard epidural placement. Ropivacaine 0.1% and Fentanyl 2mcg/mL.
  Arms: Standard Epidural (EPL)

SUMMARY:
The primary purpose of this study is to determine differences in block quality between the "dural-puncture epidural" (DPE) and standard epidural (EPL) techniques for labor analgesia in the morbidly obese patient. The investigators hypothesize that when compared to the standard EPL, the DPE technique will improve block quality .

Study participants will be randomized by computer-generated sequence to EPL or DPE arms, stratified by class of obesity (BMI 35-39.9 kg/m2, 40< 50 kg/m2 and ≥ 50 kg/m2) and by parity (nulliparous versus multiparous). All patients will receive a neuraxial technique in the sitting position at L3/4 or L4/5 using loss of resistance to saline. In the DPE group, a 25-g Whitacre needle will be used to puncture the dura. In both groups, the epidural catheter will be threaded 5 cm in the epidural space with an initiation dose of 15 ml of ropivacaine 0.1% with fentanyl (2 mcg/ml) over 6 minutes as per standard practice. After the initial loading dose and epidural pump is started, the blinded investigator will enter the patient's room to start data collection (time 0). Data will be collected for the first 30 minutes of epidural placement at 3,6,9,12,15,18 21, and 30 minutes to detect the time to achieve target pain ≤ 1/10, then assessed at standardized times (ever 2 hour) until delivery. Breakthrough pain will be managed by a standardized protocol. Other data to be collected will include: catheter adjustments and replacements, physician top-ups, asymmetrical block, pain score, motor block, sensory level to ice, hypotension, total anesthetic dose required, and PCEA use.

The primary outcome of this study is block quality defined by a composite of five components: (1) asymmetric block after 30 minutes of initiation, (2) top-up interventions, (3) catheter adjustments (4) failed catheter requiring replacement, and (5) failed epidural requiring general anesthesia or replacement neuraxial anesthesia for emergency cesarean section. Secondary outcomes include time to numeric pain rating scale ≤1, maternal adverse events (hypotension, fetal bradycardia, PDPH), motor block, duration of second stage of labor, total labor epidural time, total anesthetic dose required, PCEA use, and mode of delivery.

There is no increased risk/safety issue with placing a dural puncture technique than with epidural for labor analgesia.

DETAILED DESCRIPTION:
Purpose of the study:

The primary purpose of this study is to determine if there are differences in block quality between the DPE and standard EPL techniques for labor analgesia in the morbidly obese patient. Establishing superiority of a technique is multifaceted and complex; therefore, the design of the study will define a set of measureable outcomes to assess these properties, which will be addressed in the subsequent sections. The investigators hypothesize that when compared to the standard EPL, the DPE technique will significantly improve block quality in this population.

The secondary purpose of the study is to find an optimal maintenance regimen for epidural analgesia in the morbidly obese population. For the maintenance of epidural analgesia, it is common practice to use either continuous epidural infusion or a programmed intermittent bolus using a solution of ropivicaine 0.1% with fentanyl (2 mcg/mL). To date, there are no randomized prospective studies that investigate maintenance regimens in the morbidly obese parturient population. What has been shown is that super morbidly obese patients have increased intra-abdominal and intracranial pressure which increases pressure in the epidural space. Because of this elevated pressure, the epidural spread is increased, resulting in higher sensory blocks than necessary for adequate labor analgesia.15 An important consequence is that the morbidly obese parturient may experience additional undesirable side effects to a labor epidural: increased respiratory function, increased incidence of hypotension, and increased motor block.

Design and procedures:

The investigators propose a prospective, double-blinded, randomized trial. According to our patient population and incidence of morbid obesity, enrollment would likely occur over a 2 to 3-year period. The investigators have a delivery rate of 3500 per year. Previous data from our institution show that at least 11% of our patients are morbidly obese. The investigators will therefore expect 800-900 morbidly obese women to deliver at our institution per year. The investigators anticipate to complete enrollment for the study in 1-2 years.

Epidural technique:

Once the patient requests a labor epidural, the usual standard of care for epidural placement will be initiated. The patient will have at least one 18g intravenous catheter and will receive 500-1000 milliliter (mL) fluid administration. Vitals will be monitored by the labor nurse, including continuous pulse oximetry, non-invasive blood-pressure monitoring, and external tocodynamometry. Anesthesia time-out will be performed by the anesthesia provider with participation from the nurse and the patient.

All patients will receive a neuraxial technique in the sitting position at L3/4 or L4/5 using loss of resistance to saline. In the DPE group, a 25-g Whitacre needle will be used to puncture the dura. In both groups, the epidural catheter will be threaded 5 cm in the epidural space with an initiation dose of 15 ml of ropivacaine 0.1% with fentanyl (2 mcg/ml) over 6 minutes as per standard practice. Labor analgesia will be maintained by programmed intermittent bolus with 6 ml of the same solution every 45 minutes starting 30 minutes after the initial dose. Patients will have patient-controlled epidural analgesia (PCEA) available with an 8 ml dose per demand, every 10 minutes, for a maximum dose of 45 ml for every hour.

Assignment of Study Cohorts:

Study participants will be randomized by computer-generated sequence to EPL or DPE arms, stratified by class of obesity (BMI ≥35<40 kg/m2, ≥40<50 kg/m2 and ≥ 50 kg/m2) and by parity (nulliparous versus multiparous). Patients will be assigned to one of the four study arms by computer-generated, randomized sequence in order to balance baseline characteristics across the arms. This will be a double-blinded study. After the consented and enrolled participant requests labor epidural, a study member will give the anesthesia provider a sealed envelope with study assignment. The envelope will contain the instructions for placement of epidural with wither standard EPL or DPE technique and specified maintenance regimen of either Programmed Intermittent Epidural Bolus (PIEB) or Continuous Epidural Infusion (CEI).

Protocol for Breakthrough Pain

* If the patient has uneven or unilateral level, the provider will withdrawal catheter 1cm from skin and bolus 5ml of epidural mix. As fetal heart rate allows for maternal repositioning, the patient will lay lateral position with unblocked side in the dependent position. (up to 3 catheter adjustments)
* If the patient has bilateral levels at that below T10 to ice, the patient will be administered 5 ml off epidural pump, up to 3 times in 15 minutes.
* If the patient has pain despite T10 levels, the provider will administer Fentanyl 100 mcg via epidural.
* If analgesia continues despite these interventions up to 3 times within 30-60 minutes, the attending anesthesiologist will determine if epidural catheter needs replacement.

ELIGIBILITY:
Inclusion Criteria:

* Women admitted to the Duke Birthing Center for spontaneous or induced vaginal delivery will be screened. After usual consultation with the anesthesia team is completed and consent for anesthesia services are obtained, eligible patients will be approached to by a member of the study team.
* ages 18-45
* singleton
* vertex fetuses at 37-41 weeks' gestation
* nulliparous and multiparous women
* cervical dilation of 2-7cm
* BMI ≥ 35 kg/m2,
* pain score > 4
* English-speaking ability.

Exclusion Criteria:

* chronic opioid use
* Major cardiac disease
* contraindications to regional anesthesia

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 141 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2020-11-06 (Actual); Study Completion 2020-11-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ashraf Habib, Principal Investigator — Duke University Hospital Systems
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vricella LK, Louis JM, Mercer BM, Bolden N. Impact of morbid obesity on epidural anesthesia complications in labor. Am J Obstet Gynecol. 2011 Oct;205(4):370.e1-6. doi: 10.1016/j.ajog.2011.06.085. Epub 2011 Jun 29. PMID 21864821
- [Background] Hood DD, Dewan DM. Anesthetic and obstetric outcome in morbidly obese parturients. Anesthesiology. 1993 Dec;79(6):1210-8. doi: 10.1097/00000542-199312000-00011. PMID 8267196
- [Background] Collis RE, Davies DW, Aveling W. Randomised comparison of combined spinal-epidural and standard epidural analgesia in labour. Lancet. 1995 Jun 3;345(8962):1413-6. doi: 10.1016/s0140-6736(95)92602-x. PMID 7760614
- [Background] Cappiello E, O'Rourke N, Segal S, Tsen LC. A randomized trial of dural puncture epidural technique compared with the standard epidural technique for labor analgesia. Anesth Analg. 2008 Nov;107(5):1646-51. doi: 10.1213/ane.0b013e318184ec14. PMID 18931227
- [Background] Suzuki N, Koganemaru M, Onizuka S, Takasaki M. Dural puncture with a 26-gauge spinal needle affects spread of epidural anesthesia. Anesth Analg. 1996 May;82(5):1040-2. doi: 10.1097/00000539-199605000-00028. PMID 8610864
- [Background] Hess PE, Pratt SD, Lucas TP, Miller CG, Corbett T, Oriol N, Sarna MC. Predictors of breakthrough pain during labor epidural analgesia. Anesth Analg. 2001 Aug;93(2):414-8, 4th contents page. doi: 10.1097/00000539-200108000-00036. PMID 11473872
- [Background] Eappen S, Blinn A, Segal S. Incidence of epidural catheter replacement in parturients: a retrospective chart review. Int J Obstet Anesth. 1998 Oct;7(4):220-5. doi: 10.1016/s0959-289x(98)80042-3. PMID 15321183
- [Background] Pan PH, Bogard TD, Owen MD. Incidence and characteristics of failures in obstetric neuraxial analgesia and anesthesia: a retrospective analysis of 19,259 deliveries. Int J Obstet Anesth. 2004 Oct;13(4):227-33. doi: 10.1016/j.ijoa.2004.04.008. PMID 15477051
- [Background] Roofthooft E. Anesthesia for the morbidly obese parturient. Curr Opin Anaesthesiol. 2009 Jun;22(3):341-6. doi: 10.1097/ACO.0b013e328329a5b8. PMID 19412095
- [Background] Tien M, Allen TK, Mauritz A, Habib AS. A retrospective comparison of programmed intermittent epidural bolus with continuous epidural infusion for maintenance of labor analgesia. Curr Med Res Opin. 2016 Aug;32(8):1435-40. doi: 10.1080/03007995.2016.1181619. Epub 2016 May 20. PMID 27100210
- [Background] Gunatilake RP, Smrtka MP, Harris B, Kraus DM, Small MJ, Grotegut CA, Brown HL. Predictors of failed trial of labor among women with an extremely obese body mass index. Am J Obstet Gynecol. 2013 Dec;209(6):562.e1-5. doi: 10.1016/j.ajog.2013.07.023. Epub 2013 Jul 24. PMID 23891628
- Available data/document: Informed Consent Form: Pro00079368 — https://eirb.mc.duke.edu/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dural Puncture Epidural (DPE) | Standard Epidural (EPL)
Started | 70 | 71
Completed | 66 | 66
Not Completed | 4 | 5
Not completed — Delivered with caesarean before request for analgesia | 1 | 1
Not completed — Research staff not available | 1 | 2
Not completed — Did not receive neuraxial block | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dural Puncture Epidural (DPE) | Standard Epidural (EPL) | Total
Number analyzed (Participants) | 66 | 66 | 132
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 29.0 [25.0 to 34.0] | 30.0 [25.0 to 34.0] | 30.0 [25.0 to 34.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66 | 66 | 132
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 1 | 11
  Not Hispanic or Latino | 50 | 61 | 111
  Unknown or Not Reported | 6 | 4 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 3 | 2 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 22 | 31 | 53
  White | 26 | 26 | 52
  More than one race | 3 | 2 | 5
  Unknown or Not Reported | 10 | 5 | 15

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Required Asymmetric Block, Top-up Interventions, Catheter Adjustments, Replacement of Epidural Catheter, or Failure of Block Requiring Emergency General Anesthesia or Rescue Neuraxial Prior to Cesarean Delivery
Description: Composite outcome: asymmetric block, top-up interventions required, catheter adjustments, replacement of epidural catheter, or failure or block requiring emergency general anesthesia or rescue neuraxial prior to cesarean delivery
  Values shared are indicative of the number of participants who have the one or more of the composite elements for the composite outcome.
Time Frame: From time of randomization to time of delivery, assessed at standardized times (ever 2 hour) until delivery (estimated 72 hours).
Measure: Count of Participants; unit: Participants
Arm/Group | Dural Puncture Epidural (DPE) | Standard Epidural (EPL)
Number analyzed (Participants) | 66 | 66
Participants | 34 | 32
Statistical Analysis 1: Comparison: Dural Puncture Epidural (DPE) vs Standard Epidural (EPL); Test type: Other; p = 0.766, Regression, Logistic; Adjusted for baseline characteristics (parturient race, ethnicity, height, and induction status); Risk Difference (RD) = 3.03, 95% CI 2-sided [-14.02 to 20.08]

2. Secondary Outcome: Time to Pain Relief
Description: Time in minutes to numeric pain relief scale <= 1. Less time is better, as the pain relief scale is from 0 - 10, where 10 is the worst imaginable and 0 is no pain.
Time Frame: Data will be collected for the first 30 minutes of epidural placement to achieve target pain ≤ 1/10
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Dural Puncture Epidural (DPE) | Standard Epidural (EPL)
Number analyzed (Participants) | 66 | 66
minutes | 12 [9 to 18] | 15 [9 to 21]

3. Secondary Outcome: Degree of Motor Block as Measured by the Lowest Bromage Score
Description: The Bromage Score is used to measure degree of motor block, with a range of 1 to 5. A lower score indicates more motor block, so a higher value means a better outcome.
Time Frame: From time of randomization to time of baby delivery (estimated 72 hours)
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Dural Puncture Epidural (DPE) | Standard Epidural (EPL)
Number analyzed (Participants) | 66 | 66
score on a scale | 5 [5 to 5] | 5 [5 to 5]

4. Secondary Outcome: Number of Participants With Maternal Adverse Events
Description: Hypotension, fetal bradycardia, post-dural puncture headache
Time Frame: From time of randomization to time of 24 hours after baby delivery (estimated 72 hours)
Measure: Count of Participants; unit: Participants
Arm/Group | Dural Puncture Epidural (DPE) | Standard Epidural (EPL)
Number analyzed (Participants) | 66 | 66
Participants
  Hypotension | 2 | 6
  Fetal Bradycardia | 7 | 7
  Post-dural Puncture Headache | 0 | 0

5. Secondary Outcome: Duration of Second Stage of Labor
Description: The second stage of labor begins when the cervix is completely dilated and ends with the delivery of the baby.
Time Frame: From time of randomization to time of baby delivery (estimated 72 hours)
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Dural Puncture Epidural (DPE) | Standard Epidural (EPL)
Number analyzed (Participants) | 66 | 66
hours | 0.6 [0.16 to 1.16] | 0.32 [0.2 to 1.48]

6. Secondary Outcome: Total Labor Epidural Time
Description: Total labor epidural time
Time Frame: Total anesthetic time from time of epidural placement until discontinuation (estimated 72 hours)
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Dural Puncture Epidural (DPE) | Standard Epidural (EPL)
Number analyzed (Participants) | 66 | 66
hours | 10.76 [4.6 to 18.61] | 10.11 [6.01 to 15.19]

7. Secondary Outcome: Total Anesthetic (Ropivacaine 0.1% + Fentanyl 2) Dose Required Per Hour
Description: Consumption of epidural medications in ml including physician boluses, programmed boluses and patient controlled boluses.
Time Frame: From time of randomization to time of baby delivery (estimated 72 hours)
Measure: Median (Inter-Quartile Range); unit: mL/hour
Arm/Group | Dural Puncture Epidural (DPE) | Standard Epidural (EPL)
Number analyzed (Participants) | 66 | 66
mL/hour | 10.48 [8.54 to 14.26] | 10.88 [8.15 to 16.11]

8. Secondary Outcome: Mode of Delivery
Description: Spontaneous, assisted, or cesarean delivery
Time Frame: From time of randomization to time of baby delivery (estimated 72 hours)
Measure: Count of Participants; unit: Participants
Arm/Group | Dural Puncture Epidural (DPE) | Standard Epidural (EPL)
Number analyzed (Participants) | 66 | 66
Participants
  Spontaneous | 39 | 40
  Assisted | 4 | 3
  Cesarean delivery | 23 | 23

9. Secondary Outcome: Highest Recorded Pain Rating
Description: Numeric pain rating scale (0-10), where higher values indicate more pain or larger change.
Time Frame: From time of randomization, every 2 hours until time of delivery (estimated 72 hours)
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Dural Puncture Epidural (DPE) | Standard Epidural (EPL)
Number analyzed (Participants) | 66 | 66
score on a scale | 0 [0 to 4] | 1 [0 to 5]

10. Other Pre Specified Outcome: Satisfaction in Anesthetic Care - Likert Scale
Description: Maternal satisfaction with anesthetic care on a Likert scale from 0 - 10, 0 being unsatisfied to 10 being completely satisfied.
Time Frame: Postpartum day 1
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Dural Puncture Epidural (DPE) | Standard Epidural (EPL)
Number analyzed (Participants) | 66 | 66
score on a scale | 10 [8 to 10] | 9 [8 to 10]

ADVERSE EVENTS:
Time Frame: From time of randomization to time of 24 hours after baby delivery (estimated 72 hours)
Arm/Group | Dural Puncture Epidural (DPE) | Standard Epidural (EPL)
All-Cause Mortality (participants affected / at risk) | 0/66 | 0/66
Serious Adverse Events (participants affected / at risk) | 0/66 | 0/66
Other Adverse Events (participants affected / at risk) | 35/66 | 32/66
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dural Puncture Epidural (DPE) (N=66) | Standard Epidural (EPL) (N=66)
Hypotension (Cardiac disorders) | 2 | 6
Fetal Bradycardia (Pregnancy, puerperium and perinatal conditions) | 7 | 7
Post-dural Puncture Headache (Nervous system disorders) | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 27 | 25
Nausea (General disorders) | 11 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-16): https://cdn.clinicaltrials.gov/large-docs/95/NCT03074695/Prot_SAP_000.pdf